CLINICAL TRIAL: NCT05297123
Title: Treatment of Acute Myeloid Leukemia With Arsenic and All-trans Retinoid Acid (ATRA)
Brief Title: Treatment of Acute Myeloid Leukemia With Arsenic and All-trans Retinoid Acid
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2019LSK-077
Record Dates: First submitted 2021-10-08; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2021-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; All-trans Retinoic Acid; Arsenic
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Tretinoin; Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATRA/arsenic Group (Experimental): ATRA 20mg 3 times a day for 8 weeks Arsenic can be given intravenously (ATO) or oral Realgar-Indigo naturalis formula(RIF) ATO 0.15mg/kg/d for 8 weeks (If the total daily amount is greater than 10mg, only 10mg/d can be given) RIF 60 mg/kg/d for 8 weeks The total dose can be appropriately adjusted according to the side-effects of the drug. 4 weeks for 1 course. If the patient has obvious side effects, the treatment should stop for 2 weeks. Each patient will be received at least two courses.
  Quality of life assessments are performed every 2 months. After the end of the course of treatment, the condition is mainly evaluated based on the platelet count and bone marrow smear. If the treatment is effective, the above regimen can be continued; if not, the study is withdrawn.
  Interventions: Drug: All-trans retinoic acid; Drug: Arsenic Trioxide; Drug: Realgar-Indigo naturalis formula

INTERVENTIONS:
Drug: All-trans retinoic acid — All-trans retinoic acid (ATRA) 20mg 3 times a day for 8 weeks.
  Other Names: ATRA
Drug: Arsenic Trioxide — ATO 0.15mg/kg/d for 8 weeks (If the total daily amount is greater than 10mg, only 10mg/d can be given)
  Other Names: ATO
Drug: Realgar-Indigo naturalis formula — 60 mg/kg/d for 8 weeks
  Other Names: RIF

SUMMARY:
The clinical trial was designed to prove that Arsenic plus ATRA possibly had an effect on improving the symptoms, reducing the early mortality rate and prolonging the total survival time of patients with newly diagnosed or relapsed AML.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a genetically heterogeneous disease with a highly variable prognosis and an overall high mortality rate. The 5-year overall survival of adult AML patients is less than 50%, and only 20% of elderly patients survive over 2 years. Acute promyelocytic leukemia (APL) accounts for 10% - 15% of acute myeloid leukemia. Arsenic and ATRA are very effective treatments for APL, a distinct AML subtype characterized by the expression of the PML/RARA fusion protein. PML/RARA expression disrupts PML NBs and blunts p53 signaling, which contributes to increased self-renewal of myeloid progenitors. The application of all-trans retinoic acid (ATRA) and arsenic modifies APL from highly fatal to highly curable. Both RA and arsenic induce degradation of PML/RARA through distinct pathways. Nucleophosmin-1(NPM1) is the most frequently mutated gene in acute myeloid leukemia (AML). According to El Hajj's research, RA or arsenic trioxide synergistically induces proteasomal degradation of mutant NPM1 in AML cell lines or primary samples, leading to differentiation and apoptosis. Combined ATRA/arsenic treatment significantly reduced bone marrow blasts in 3 AML patients and restored the subnuclear localization of both NPM1 and PML. Overall, there is no consensus yet as to whether the addition of ATRA/arsenic improves the outcome of patients with NPM1 mutant AML. However, it still needs clinical research to confirm. The investigators design a clinical trial to prove that arsenic plus ATRA is possibly improving the symptoms of AML patients, reduce early mortality, and extending overall survival time.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or relapsed AML.Diagnosis based on Chinese guidelines for diagnosis and treatment of adult acute myeloid leukemia(not APL)(2018)
* Older than 18 years old
* Patients or their families signed written informed consent

Exclusion Criteria:

* Be allergic to the drug ingredient, the supplementary material or the allergic constitution person
* Cardiac insufficiency, renal insufficiency, significant arrhythmias, EKG abnormalities or other important organ dysfunction
* Combined with other malignant tumors
* Pregnant and lactating women
* Participants in other drug trials in the last 3 months
* Suffering from mental illness or other circumstances which unable to carry out the plan
* Other patients who were not suitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-03 (Actual); Primary Completion 2023-12-03 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Early death rate (ED) | 30 days
  Death reported within the first month of diagnosis
Overall survival (OS) | From date of enrollment until the date of death from any cause, assessed up to 3 years
  the time from enrolled to death from any cause

SECONDARY OUTCOMES:
Hematologic complete remission (HCR) | 30 days
  Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0×10^9 /L; platelet count >100× 10^9 /L.
Cumulative relapse rate | From the date of enrollment to the date of relpase proved by bone marrow test, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Huaiyu Wang, Dr., Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennett DA. How can I deal with missing data in my study? Aust N Z J Public Health. 2001 Oct;25(5):464-9. PMID 11688629
- [Background] Dos Santos GA, Kats L, Pandolfi PP. Synergy against PML-RARa: targeting transcription, proteolysis, differentiation, and self-renewal in acute promyelocytic leukemia. J Exp Med. 2013 Dec 16;210(13):2793-802. doi: 10.1084/jem.20131121. PMID 24344243
- [Background] de The H, Chen Z. Acute promyelocytic leukaemia: novel insights into the mechanisms of cure. Nat Rev Cancer. 2010 Nov;10(11):775-83. doi: 10.1038/nrc2943. Epub 2010 Oct 22. PMID 20966922
- [Background] Zhao Z, Zuber J, Diaz-Flores E, Lintault L, Kogan SC, Shannon K, Lowe SW. p53 loss promotes acute myeloid leukemia by enabling aberrant self-renewal. Genes Dev. 2010 Jul 1;24(13):1389-402. doi: 10.1101/gad.1940710. PMID 20595231
- [Background] El Hajj H, Dassouki Z, Berthier C, Raffoux E, Ades L, Legrand O, Hleihel R, Sahin U, Tawil N, Salameh A, Zibara K, Darwiche N, Mohty M, Dombret H, Fenaux P, de The H, Bazarbachi A. Retinoic acid and arsenic trioxide trigger degradation of mutated NPM1, resulting in apoptosis of AML cells. Blood. 2015 May 28;125(22):3447-54. doi: 10.1182/blood-2014-11-612416. Epub 2015 Mar 23. PMID 25800051